CLINICAL TRIAL: NCT04322448
Title: Identification and Validation of Non-invasive Mechanomyography as a Valuable Predictor of Clinical Course and Long-term Prognosis for Cubital Tunnel Syndrome and Peroneal Nerve Decompression Patients
Brief Title: Mechanomyography for Predictor of Prognosis in CuTS and PND Patients
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Wilson Z. Ray, Principal Investigator, Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Other Study IDs: 201905017
Record Dates: First submitted 2020-01-27; First posted 2020-03-26 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2024-11

CONDITIONS: Cubital Tunnel Syndrome; Peroneal Nerve Entrapment
Keywords: cubital tunnel; cubital; peroneal; nerve entrapment; nerve compression; nerve decompression; CuTS; PND; MMG; mechanomyography; cubital tunnel syndrome; peroneal nerve decompression
MeSH Terms: conditions — Cubital Tunnel Syndrome; Peroneal Neuropathies; Nerve Compression Syndromes; Neuroma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Cubital Tunnel Syndrome Patients: Cubital Tunnel Syndrome patients. Patients will undergo standard of care exams and surgery. During surgery, the surgeon will apply the mechanomyography (MMG) to the targeted nerve immediately prior and post decompression. Subjects will be followed until they are 6 months postop.
  Interventions: Device: Mechanomyography (MMG)
- Peroneal Nerve Decompression Patients: Patients with compressive peroneal nerve neuropathy and will undergo a Peroneal Nerve Decompression (PND). Patients will undergo standard of care exams and surgery. During surgery, the surgeon will apply the mechanomyography (MMG) to the targeted nerve immediately prior and post decompression. Subjects will be followed until they are 6 months postop.
  Interventions: Device: Mechanomyography (MMG)

INTERVENTIONS:
Device: Mechanomyography (MMG) — MMG, as described in the cohort descriptions, to be used during surgery to see if they are predictive of patient outcomes.

SUMMARY:
The study will be a non-blinded two cohort design consisting only of symptomatic patients with CuTS or compressive peroneal neuropathy or in need of peroneal nerve decompression. The first cohort will be - patients with CuTS. Evaluation of each CuTS patient will include assessment by the treating surgeon and a certified hand therapist. Patients who have clinical examination and history consistent with a diagnosis of CuTS based on subjective and functional assessment outlined below will be consented to this study. The second cohort will be patients in need PND for compressive neuropathy of peroneal nerve. PND patients will be evaluated by clinical exam and have imaging with high resolution ultrasound or MRI negative for mass lesion.

DETAILED DESCRIPTION:
Visit 1

* Exam and discussion with surgeon
* Exam and testing with Occupational Hand Therapist (Standard of Care) as described above. (CuTS cohort)
* Diagnostic studies (EMG/NCT) (Standard of Care)
* Questionnaires - PROMIS and ODI

Visit 2

* Standard of Care surgery
* During surgery, the surgeon will perform an MMG immediately pre-decompression and immediately post-decompression of the nerve. This will entail placing a sensor and probe on the nerve that will be decompressed.

Visit 3 and 4 (6 week and 3 month post-op)

* Clinical Exam by Surgeon
* Exam and testing with Occupational Therapist (Standard of Care) as described above. (CuTS cohort)
* Questionnaires - PROMIS and ODI

Visit 5 (6 months post-op)

* Clinical Exam by Surgeon
* Exam and testing with Occupational Therapist (Standard of Care) as described above. (CuTS cohort)
* Questionnaires - PROMIS and ODI
* Evaluation of MMG parameters

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a diagnosis of Cubital Tunnel Syndrome or Compressive Peroneal Nerve Neuropathy and will be undergoing a decompressive surgery.

Exclusion Criteria:

* Patients under 18 years of age
* Patients who are unable to return for follow-up evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited in the investigator's patient population.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
PROMIS Questionnaire | 6 months
  PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. Scores range from 0-50 with a higher indicating a better outcome.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | 6 months
  10 question tool that researchers and disability evaluators use to measure a patient's permanent functional disability. Score ranges from 0-100. Lower scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Z Ray, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No